CLINICAL TRIAL: NCT00494884
Title: A Multicenter, Randomized, Double-blind, Parallel-group Study to Investigate the Glucose Lowering Effect, Safety and Tolerability of 24 Weeks Treatment With Vildagliptin 100 mg o.d. Versus Placebo Followed by a 12 Weeks Treatment Period With Open-label Vildagliptin 100 mg o.d. as add-on Therapy in Patients With Type 2 Diabetes Inadequately Controlled With Metformin
Brief Title: Vildagliptin 100 mg Once Daily vs. Placebo as add-on Therapy in Patients With Type 2 Diabetes Inadequately Controlled With Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237ADE02
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin; metformin combination
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
This study will investigate efficacy and safety of vildagliptin in patients with low baseline levels starting at an HbA1C level of 6.5% to support convenient early intervention with combination therapies. In parallel, morning and evening dosing will be evaluated in this patient population for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Male, non-fertile female or female of childbearing potential using a medically approved birth control method
* Patients who have received metformin for at least three months prior to visit 1 and have been on a stable dose for a minimum of 8 weeks prior to visit 1
* Agreement to maintain the same dose of metformin throughout the study
* Age in the range of 18-85 years inclusive.
* HbA1c in the range of 6.5 - 8.0% (inclusive) at visit 1
* Agreement to maintain prior diet and exercise habits during the full course of the study
* Ability to comply with all study requirements and signed informed consent to participate in the study.

Exclusion Criteria:

* Pregnant or lactating female

A history of:

* type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes, e.g. Cushing's syndrome and acromegaly.
* acute metabolic diabetic complications such as ketoacidosis or hyperosmolar state (coma) within the past 6 months.

Any of the following significant laboratory abnormalities:

* ALT, AST greater than 2 times the upper limit of the normal range at visit 1.
* Direct bilirubin greater than the upper limit of the normal range at visit 1.
* Serum creatinine levels equal to or greater than 1.5 mg/dL (132 umol/L) males, equal to or greater than 1.4 mg/dL (123 umol/L) females, or a history of abnormal creatinine clearance at visit 1.
* Clinically significant TSH values outside of normal range at visit 1.
* Clinically significant laboratory abnormalities, confirmed by repeat measurement, other than hyperglycemia, hyperinsulinemia, and glycosuria at visit 1 Treatment with any oral anti-diabetic other than metformin within 3 months prior to visit 1

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose | 24 weeks
Adverse event profiles including gastrointestinal tolerability and hypoglycemia | 24 weeks
Responder rates | 24 weeks
Change from baseline in insulin and proinsulin in a subgroup of patients | 24 weeks
Change in systolic and diastolic blood pressure | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. W. E. Schmidt, Study Director — Ruhr-Universitat Bochum, Medizinische Klinik, St. Josef Hospital, Gudrunstr. 56, D-44791 Bochum, Telefon: 0234-509-2311, Telefax: 0234-509-2309
Locations (1):
- Novartis Investigative Site, Bochum, Germany